CLINICAL TRIAL: NCT06216873
Title: Collecting the Results of Physical Examination, Blood Test, and Radiological Examination of Multiple Trauma Patients With Activated Trauma Team and Understanding the Correlation With Patient's Morality and Mobility
Brief Title: Collecting the Results of Multiple Trauma Patients and Find the Correlation of Morality and Mobility
Acronym: trauma
Status: Recruiting | Type: Observational
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Principal Investigator, Chia-hsi Chen, Physician of Emergency Medicine, St. Martin De Porress Hospital
Other Study IDs: 23B-021
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Multiple Trauma/Injuries
Keywords: Trauma; physical parameter; radiologic examination
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple trauma: multiple trauma patients sent to emergency room for further evaluation are included
  Interventions: Other: multiple trauma

INTERVENTIONS:
Other: multiple trauma — Review the medical record to gather the physical parameters, blood examination result and radiologic examination results

SUMMARY:
Collect data about physiological examination values, blood test values and radiological examination results of patients admitted to the hospital for major trauma. There are different causes of mortality in multiple trauma patients. In this study, review the multiple symptoms and parameters of major trauma patients. We hope to understand and develop one feasible assessment model for emergency departments for enable rapid diagnosis and treatment evaluation about major trauma patients occurrence.

DETAILED DESCRIPTION:
1. This is a retrospective study of patients admitted to the emergency department at a single center, focusing on reviewing their medical records and patient examination performance.
2. The parameters including hospital on-site records and patient examination result, physiological examination values, blood test values and radiological examination results.on the medical records of patients who visited emergency department are collected.
3. This study will explore how to improve the response and effectiveness of investigating patients when they are admitted to the hospital for major trauma.
4. Evaluate the effectiveness and efficiency of this operative model to increase the possibility of receiving medical examination, timely correct diagnosis on major trauma patients when they sent to the emergency department, and improve the hospital's manpower deployment plan.

ELIGIBILITY:
Inclusion Criteria:multiple trauma patients -

Exclusion Criteria:expired patients at emergency room

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The multiple trauma patients are sent to emergency room for further evaluation and management.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The Survey of Mortality and Mobility on Multiple Trauma Patients | 20100101 till 20260731
  Analyze and evaluate the effectiveness of this operative model to increase the possibility of correct diagnosis and timely medical examination major trauma patients and improve the hospital's manpower deployment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Chia Hsi Chen, MD, Principal Investigator — Department of Emergency, St. Martin De Porres Hospital
Locations (1):
- St. Martin De Porres Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The individual participant data include the personal medical data and should not be shared with other researchers.